CLINICAL TRIAL: NCT05164250
Title: Compassionate Use (CU) of REGN5458 for Patients With Relapsed or Refractory Multiple Myeloma (MM)
Status: Approved for marketing | Type: Expanded Access
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: R5458-MM
Record Dates: First submitted 2021-12-09; First posted 2021-12-20 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-10

CONDITIONS: Multiple Myeloma
Keywords: Relapsed, Refractory
MeSH Terms: conditions — Multiple Myeloma; Recurrence

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: REGN5458
  Other Names: BCMAxCD3; linvoseltamab

SUMMARY:
Provide Compassionate Use' of REGN5458 for Patients with Relapsed or Refractory Multiple Myeloma

DETAILED DESCRIPTION:
Compassionate Use requests are only being considered in response to Individual Patient Investigational New Drug (IND) applications.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

-

Age Groups: Child, Adult, Older Adult